CLINICAL TRIAL: NCT00394992
Title: Randomized Phase III Study Post Radical Resection of Liver Metastasis of Colorectal Cancer: Bevacizumab in Combination With XELOX as Adjuvant Chemotherapy vs XELOX Alone
Brief Title: Adjuvant Xeloda Plus Eloxatin +/- Avastin After Radical Resection of Liver Metastasis of Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data from the C08 study and Avant study
Sponsor: Dutch Colorectal Cancer Group (Other)
Collaborators: Sanofi (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPATICA
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Colorectal cancer; Liver metastasis; Radical resection; Adjuvant therapy; Bevacizumab; Capecitabine; Oxaliplatin; Hepatica
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 oxaliplatin+capecitabine (Active Comparator): postoperatively oxaliplatin 130 mg/m2 i.v. day 1 plus capecitabine 1000 mg/m2 b.i.d. on day 1-14, q3w
  Interventions: Drug: oxaliplatin+capecitabine
- 2 oxaliplatin+capecitabine+bevacizumab (Experimental): postoperatively oxaliplatin 130 mg/m2 i.v. day 1 plus bevacizumab 7.5 mg/kg on day 1 plus capecitabine 1000 mg/m2 b.i.d. on day 1-14, q3w
  Interventions: Drug: Oxaliplatin+capecitabine+bevacizumab

INTERVENTIONS:
Drug: oxaliplatin+capecitabine — postoperatively oxaliplatin 130 mg/m2 i.v. day 1 plus capecitabine 1000 mg/m2 b.i.d. on day 1-14, q3w
  Arms: 1 oxaliplatin+capecitabine
Drug: Oxaliplatin+capecitabine+bevacizumab — postoperatively oxaliplatin 130 mg/m2 i.v. day 1 plus bevacizumab 7.5 mg/kg on day 1 plus capecitabine 1000 mg/m2 b.i.d. on day 1-14, q3w
  Arms: 2 oxaliplatin+capecitabine+bevacizumab

SUMMARY:
The primary aim of this study is to investigate whether the addition of the new anti-cancer drug bevacizumab (Avastin) to the combination of the chemotherapeutic agents capecitabine (Xeloda) and oxaliplatin (Eloxatin) reduces (slows down) the recurrence of metastatic disease after a radical resection of liver metastases in patients with colorectal cancer.

DETAILED DESCRIPTION:
The primary therapy of colorectal cancer is surgical resection, but more than half of all colorectal cancer patients eventually die of metastatic disease. Although the introduction of new anticancer agents with efficacy in metastatic colorectal cancer, e.g.: oxaliplatin and irinotecan, and the targeted agents cetuximab and bevacizumab has changed therapeutic nihilism, chemotherapy alone has failed to cure these patients.

It is estimated that 15-20 % of colorectal cancer patients present with synchronous liver metastases and approximately 50% of the patients with colorectal tumors will develop liver metastases at some point during the course of their disease. In almost one third of the cases, the liver was shown at autopsy to be the only site of cancer spread. This is in accordance with the 20% - 45 % five-year survival obtained with surgical resection of hepatic metastases.

Previous studies have not shown a clear benefit of adjuvant chemotherapy after metastasectomy of liver metastases. However, most of these studies have been performed with 5-fluorouracil with or without other older cytostatic drugs. Since new effective agents have been developed (e.g.: capecitabine, oxaliplatin and bevacizumab), adjuvant combination treatment with these agents might be more effective. These drugs have proven activity as first line palliative treatment of recurrent metastases. This raises the question if this new effective treatment is of value as an adjuvant treatment after metastasectomy.

As mentioned before, a two-arm EORTC study: neoadjuvant and adjuvant FOLFOX vs no chemotherapy in resectable liver metastases of colorectal cancer is almost completed (Nordlinger et al). It is expected that this study will show a 10% 3 year DFS benefit in favour of th treatment arm. Definitive data of this trial will be released at the end of 2006, and will most probably lead to adjuvant treatment post metastasectomy as a standard of care. In the HEPATCIA trial we anticipate on this by using adjuvant XELOX as the control arm.

As mentioned earlier, the 3-year disease free survival in patients post metastasectomy of liver metastases is approximately 25%. There is no data available on the effectivity of the XELOX regimen as adjuvant treatment after metastasectomy of colorectal cancer metastases. The EORTC study was designed to demonstrate a 10% improvement in 3y DFS. Assuming that this study is positive, 3 year DFS would be 35% in the control arm (XELOX post liver resection).

Since bevacizumab inhibits angiogenesis, which is required for growth of metastases, this drug may be valuable in the adjuvant setting. Several studies investigate the value of this drug in combination with fluoropyrimidines as an adjuvant regimen after resection of primary colorectal cancers. However, at this moment there is no mature data available of these studies. Therefore, we assume an increase in 3-year disease free survival of 10%, to 45% in the XELOX and bevacizumab treatment arm.

This study will therefore evaluate patients with resectable liver metastasis without extra-hepatic disease, investigating whether the capecitabine, oxaliplatin and bevacizumab regimen is superior to capecitabine and oxaliplatin alone applied as adjuvant treatment, in order to extent disease free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to any study-specific procedures.
* Age ≥ 18 years.
* Liver metastases radically resected (R0 resection).
* Study medication started ≥4 and ≤ 8 weeks post liver surgery.
* Histologically confirmed liver metastasis of colorectal cancer after surgery.
* ECOG performance status 0 or 1.
* Adequate hematology: ANC ≥1.5 x 109/L, platelets ≥100 x 109/L, Hb ≥5.5 mmol/L, INR ≤ 1.5, APTT < 1.5 X UNL.
* Adequate biochemistry: total bilirubin ≤1.5 UNL, ASAT and ALAT ≤2.5 x UNL, alkaline phosphatase ≤2.5 x UNL, serum creatinine ≤1.5 UNL.
* Urine dipstick <2+ for protein.

Exclusion Criteria:

* Extrahepatic metastatic disease.
* Prior adjuvant chemotherapy given <6 months prior to detection of the liver metastases.
* Prior non colorectal malignancies.
* Bleeding diathesis or coagulation disorders or the need for full-dose anticoagulation.
* Major surgical procedure <4 weeks prior to start of study treatment.
* Females with a positive pregnancy test (within 14 days before treatment start) .
* Lactating women.
* Fertile women (<2 years after last menstruation) and women of childbearing potential not willing to use effective means of contraception.
* History of psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant (i.e. active) cardiovascular disease e.g. cerebrovascular accidents (≤6 months prior to randomization), myocardial infarction (≤1 year prior to randomization), uncontrolled hypertension while receiving chronic medication, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Known peripheral neuropathy, including oxaliplatin induced neuropathy > grade Absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible.
* Organ allografts requiring immunosuppressive therapy.
* Serious, non-healing wound, ulcer, or bone fracture.
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes.
* Chronic, daily treatment with high-dose asprin (> 325 mg/day) or nonsteroidal anti-inflammatory medications (those known to inhibit platelet function at doses used to treat chronic inflammatory diseases). Patients can be rendered eligible by changing the treatment to COX II inhibitors.
* Chronic treatment with corticosteroids (dose of ≥ 10 mg/day methylprednisolone equivalent excluding inhaled steroids).
* Serious intercurrent infections (uncontrolled or requiring treatment).
* Current or recent (within the 28 days prior to randomization) treatment with another investigational drug or participation in another investigational study.
* Patients with known allergy to Chinese hamster Ovary cell proteins or other recombinant human or humanized antibodies or to any excipients of bevacizumab formulation, platinum compounds or to any other component of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
3-year disease free survival, defined as the percentage of disease free patients 3 year after randomisation. | study duration

SECONDARY OUTCOMES:
Overall survival, defined as the percentage of patients alive 5 year after randomisation. | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Richard van Hillegersberg, MD PhD, Principal Investigator — Universitair Medisch Centrum Utrecht
Locations (1):
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Snoeren N, Voest EE, Bergman AM, Dalesio O, Verheul HM, Tollenaar RA, van der Sijp JR, Schouten SB, Rinkes IH, van Hillegersberg R. A randomized two arm phase III study in patients post radical resection of liver metastases of colorectal cancer to investigate bevacizumab in combination with capecitabine plus oxaliplatin (CAPOX) vs CAPOX alone as adjuvant treatment. BMC Cancer. 2010 Oct 11;10:545. doi: 10.1186/1471-2407-10-545. PMID 20937118
- See also: Websites Dutch Colorectal Cancer Group — http://www.dccg.nl
- See also: University Medical Center Utrecht — http://www.umcutrecht.nl/research/